CLINICAL TRIAL: NCT06036082
Title: Improvement by Isokinetic and Treadmill Training on Muscle Strength and Gait in Burned Children
Brief Title: Isokinetic Training Versus Treadmill Training on Muscle Strength and Gait in Children With Lower Limb Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ragaee Saeed Mahmoud, Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/2111/MTI.PT/2204062
Record Dates: First submitted 2023-09-02; First posted 2023-09-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Burned
Keywords: Burn; Children; Isokinetic Training; Treadmill Training
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: randomized control study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional physical therapy group (Experimental): It consisted of 20 children received conventional physical therapy program
  Interventions: Other: Conventional physical therapy
- isokinetic training group (Experimental): It consisted of 20 children received conventional physical therapy program and isokinetic training
  Interventions: Other: Conventional physical therapy
- Treadmill training group (Experimental): It consisted of 20 children received conventional physical therapy program and treadmill training
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Conventional physical therapy — * Standing with feet together .
  * Step standing .
  * High step standing and trying to keep balanced.
  * Single leg stance "unilateral standing" with assistance.
  * Standing on a declined surface by using wedge.
  * Standing with manual locking of the knees.
  * Changing position.
  * Gait training.
  * Static and dynamic muscle contraction.
  Other Names: physical therapy program

SUMMARY:
Burn wounds are one of the most complexes and dramatic of all injuries, it produces a direct local tissue destruction and damage. In addition, burn wounds may continue to destroy tissue and muscles, exercise therapy stimulates the early expression of angiogenesis-related growth factors so it results in new vessel in-growth that improves blood supply, increases cell proliferation, accelerates tissue regeneration and healing and regain muscle strength

DETAILED DESCRIPTION:
To evaluate the efficacy of isokinetic training against treadmill training in improving muscle strength and gait in children having lower limb burns. Methods: Sixty children from both genders (boys and girls) who were complaining from 2nd degree lower limb burns with ≥30 percent of their total body surface area (TBSA) participated in this study, their ages ranged from 8 to 16 years and they were randomized into three groups of same number (A, B and C). Groups (A) received conventional physical therapy program, group (B) received the same conventional physical therapy program of group (A) with trained to use the isokinetic device while group (C) received the same conventional physical therapy program of group (A and B) and used treadmill training. The children participated in this study were assessed by Hand-held dynamometer (HHD) and Balance Master System (BMS). They were evaluated before and after the treatment program three sessions per week for 12 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8 to 16 year
* Complaining from 2nd degree lower limb burns (≥30 % of their TBSA).
* Capable of standing and walking independently.
* Clinically and medically stable.
* Sufficient cognition demonstrating understanding the requirements of the study.
* No history of lower extremity surgery.

Exclusion Criteria:

* Visual and/or auditory defects.
* Significant shortening and/or deformity of lower extremities.
* Other neurological problems that affect balance or mentality (e.g. epilepsy).
* Advanced radiographic changes include (bone destruction, bony ankylosis, knee joint sublaxation and epiphysial fracture).
* Congenital or acquired skeletal deformities in the lower limbs.
* Cardiopulmonary dysfunction.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Balance Master System | before intervention and after 12 weeks of intervention
  It is the most significant test to measure balance and has valid values of functional balance performance

SECONDARY OUTCOMES:
Hand-held dynamometer | before intervention and after 12 weeks of intervention
  It is a portable device (Nicholas Manual Muscle Tester, Model 01160; Lafayette Instrument, Lafayette, IN), characterized as low-cost and convenient method

CONTACTS AND LOCATIONS:
Locations (1):
- Ragaee Saeed Mahmoud, Faisal, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
assessed before and after treatment
Supporting Information: Study Protocol
Time Frame: 12 weeks
Access Criteria: accepted